CLINICAL TRIAL: NCT03788824
Title: Evaluation of Inflammation Activity in Ulcerative Colitis by Probe-based Confocal Laser Endomicroscopy
Brief Title: Evaluation of Inflammation Activity in Ulcerative Colitis by pCLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2014SDU-QILU-G05
Record Dates: First submitted 2014-11-13; First posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Inflammation
Keywords: Ulcerative Colitis; probe-based Confocal Laser Endoscopy; Inflammation Activity; Histology
MeSH Terms: conditions — Inflammation; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sample for histological examination
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pCLE group: pCLE is used to distinguish the inflammation activity of UC, and compared with histology

SUMMARY:
The aim:1) To test the correlation of pCLE-obtained features with histological findings in UC; comparing the real-time conventional colonoscopy Baron score with CLE assessment. 2) To test the accuracy of the investigators previously proposed simplified four-grade classification system of crypt architecture in evaluating inflammation activity in UC by pCLE.

DETAILED DESCRIPTION:
Patients with acute inflammatory infiltrates seen on histological assessment are more likely to experience relapse than are those without infiltrates,studies suggest that severity of inflammation is a risk factor for colorectal neoplasia in UC.

The assessment of inflammation activity by conventional colonoscopy is inaccurate in the prediction of acute inflammation in some cases. Confocal laser endomicroscopy (CLE) allows for real-time endoscopy and histological diagnosis of gastrointestinal diseases. In our previous study, we confirmed a simplified four-grade classification system of crypt architecture(Grade A :normal; Grade B: an irregular arrangement of colonic crypts with normal size and shape, and enlarged spaces between crypts; Type C: an enlarged crypt opening and a more irregular crypt arrangement than type B; Type D: crypt destruction and / or crypt abscess) by eCLE in predicting acute inflammation, and found a good correlation with histology. In this study, the investigators aimed to test the accuracy of the proposed tne four-grade classification system in evaluating inflammation activity in UC by pCLE.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 18-80;
* patients previously or in-process diagnosed as Ulcerative Colitis

Exclusion Criteria:

* Patients with gastrectomy, acute GI bleeding, and advanced esophageal cancer;
* Patients under conditions unsuitable for performing CLE including coagulopathy (prothrombin time <50% of control, partial thromboplastin time >50 s), lactation, food retention, oesophageal stenosis, postoperative cases, leiomyoma, impaired renal function (creatinine level >1.2 mg/dL), pregnancy or breastfeeding, and known allergy to fluorescein sodium;
* Inability to provide informed consent and other situations that could interfere with the examination protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients screened that fulfill the eligibility criteria at Qilu Hospital, Shandong University will be enrolled into the study
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
A valuable realtime- and offline- diagnosis of pCLE in evaluating the inflammation activity in UC. | 2 years
  Recruited more than 100 UC patients,pCLE diagnostic criteria was the four-grades crypt architecture classification system ( inactive cases with Grade A or B, active with Grade C or D), histological assessment according to the Geboes Index ( inactive disease with Geboes index ≤ 3.0; active disease with a index > 3.0). Using Spearman's text, calculating the corelation between pCLE real-time finding and the Geboes index, if p<0.05, it means a strong corelation,vice versa. Also for the offline diagnosis.
  Also calculate the corelation between white-light colonoscopy (Baron Score) and histopathology.

SECONDARY OUTCOMES:
Good or Excellent interobserver and intraobserver agreement of pCLE diagnosis. | 2 years
  Assessment of interobserver variability of pCLE was conducted in a randomized pCLE videos' order by two independent investigators. After a 2-week interval, all pCLE videos were reassessed by the two investigators to evaluate the intraobserver agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD. PhD., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China